CLINICAL TRIAL: NCT01133730
Title: The Analgesic Efficacy of the Transversalis Fascia Plane Block in Iliac Crest Bone Graft Harvesting
Brief Title: Transversalis Fascial Plane Nerve Block in Iliac Crest Bone Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-0200-A
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2010-05

CONDITIONS: Upper Limb Surgery; Iliac Crest Bone Harvest
Keywords: supraclavicular nerve block; regional anesthesia; transversalis fascia plane block; ultrasound guided; opioid consumption; iliac crest bone harvest; hand surgery; wrist surgery; Upper limb surgery combined with iliac crest bone harvest.

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active treatment group (Experimental): Ultrasound-guided TFP block with 20ml 0.5% ropivacaine + 1:200 000 epinephrine
  Interventions: Drug: Active treatment
- Placebo arm (Placebo Comparator): Ultrasound-guided TFP block with 20ml of 5% dextrose solution
  Interventions: Drug: Placebo Arm

INTERVENTIONS:
Drug: Active treatment — US-guided TFP block with 20ml 0.5% ropivacaine + 1:200 000 epinephrine
  Arms: Active treatment group
Drug: Placebo Arm — US-guided TFP block with 20ml of 5% dextrose solution
  Arms: Placebo arm

SUMMARY:
Hand or wrist surgery often requires the use of bony material in order to accomplish any associated reconstructive aspects required for the surgery. The iliac crest is often used as the source of bone for such surgery and harvesting from this site is performed simultaneously with the hand/wrist surgery. In terms of anesthesia, patients typically receive a supraclavicular nerve block for the hand/wrist surgery, and a general anesthestic for the bone graft, though spinal block may also be performed. This study will look at the use of a transversalis fascia plane (TFP) nerve block (ie, to numb the nerves going to the iliac crest) in combination with a general anesthetic to see if post-operative pain and opioid consumption is reduced using the TFP block.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I-III
2. 18-85 years of age, inclusive
3. Weight 50kg+
4. Scheduled for elective upper limb surgery, which can be solely performed under a brachial plexus block, and requiring an ICBG

Exclusion Criteria:

1. Contraindications to regional blockade (e.g., allergy to local anesthetics, coagulopathy, malignancy or infection in the area)
2. Pregnancy
3. History of alcohol or drug dependency/abuse
4. History of long term opioid intake or chronic pain disorder
5. History of significant psychiatric conditions that may affect patient assessment
6. Failure of upper extremity block
7. Previous iliac crest bone grafting
8. History of severe pelvic and hip conditions that could interfere with the long-term functional assessments of the study
9. Inability to understand the informed consent and demands of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 24 hours
  Opioid consumption in the first 24 hours following ICBG. This will be expressed in terms of milligrams doses of IV morphine. Where other opioids are used, the doses will be converted to the equivalent IV morphine dose using standard opioid dosage conversion tables.

SECONDARY OUTCOMES:
Opioid consumption | 7 days
  Opioid consumption (expressed as milligram doses of IV morphine) in the following phases
  * Intraoperative phase (from start of surgery to end of surgery)
  * Postoperative care unit stay (from admission to discharge)
  * First 48 hours following ICBG
Pain measures | 48 hours
  * Pain scores at the ICBG site, measured using a visual analogue scale (VAS) (scale 0-10) and starting in recovery, then every 4 hrs for the next 48 hrs.
  * Pain at the primary surgical site (VAS 0-10)
  * Duration of block, defined as the time from completion of block performance to the time of onset of increased pain at the ICBG harvest site (as perceived by the patient)
Time of block performance | 6 hours
  Time required to perform the TFP block (defined as the time between placement of the ultrasound probe on the patient, and withdrawal of the block needle)
Complications | 12 months
  TFP block complications and adverse events (e.g. vascular puncture, intravascular local anesthetic injection and local hematoma)

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada